CLINICAL TRIAL: NCT04639414
Title: Combined Active Treatment in Type 2 Diabetes with NASH
Acronym: COMBAT_T2_NASH
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: German Diabetes Center (Other)
Collaborators: Boehringer Ingelheim (Industry); German Center for Diabetes Research (Other); Federal Ministry of Health, Germany (Other Government); Ministry of Innovation, Science and Research in North Rhine-Westphalia (Unknown); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Combat_T2_NASH_002; 2019-001987-31 (EudraCT Number)
Record Dates: First submitted 2019-04-05; First posted 2020-11-20 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes; Non-alcoholic Steatohepatitis (NASH); Non-alcoholic Fatty Liver Disease (NAFLD)
Keywords: Type 2 Diabetes; Non-alcoholic Steatohepatitis (NASH); Non-alcoholic Fatty Liver Disease (NAFLD); Fatty liver; Diabetes mellitus; Empagliflozin; Semaglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Fatty Liver; Diabetes Mellitus | interventions — empagliflozin; Tablets; semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Combined treatment with Empagliflozin and Semaglutide (Experimental): Combined treatment with Empagliflozin, film-coated tablet, 10mg once daily and Semaglutide, colourless solution in pre-filled pen, 1mg once weekly
  Interventions: Drug: Empagliflozin 10mg oral tablet / Semaglutide 1mg pen injector
- Empagliflozin monotherapy (Experimental): Empagliflozin, film-coated tablet, 10mg once daily and Placebo matching Semaglutide (colourless solution in pre-filled pen, once weekly)
  Interventions: Drug: Empagliflozin 10mg oral tablet and placebo pen injector matching semaglutide
- Placebo (Placebo Comparator): Placebo matching Empagliflozin (film-coated tablet, once daily) and Placebo matching Semaglutide (colourless solution in pre-filled pen, once weekly)
  Interventions: Drug: Placebo matching empagliflozin and placebo pen injector matching semaglutide

INTERVENTIONS:
Drug: Empagliflozin 10mg oral tablet / Semaglutide 1mg pen injector — Measurement of the effect of the combined treatment with semaglutide 1mg/week and empagliflozin 10 mg/d compared to matching placebo after 48-week treatment.
  Other Names: Jardiance(R), Ozempic(R)
  Arms: Combined treatment with Empagliflozin and Semaglutide
Drug: Empagliflozin 10mg oral tablet and placebo pen injector matching semaglutide — Measurement of the effect of empagliflozin monotherapy 10mg/d compared to matching placebo after 48-week treatment.
  Other Names: Jardiance(R)
  Arms: Empagliflozin monotherapy
Drug: Placebo matching empagliflozin and placebo pen injector matching semaglutide — Measurement of the effect of the combined treatment with semaglutide 1mg/week and empagliflozin 10 mg/d OR empagliflozin monotherapy 10mg/d compared to matching placebo after 48-week treatment.
  Other Names: Control / Placebo
  Arms: Placebo

SUMMARY:
The aim of this multicentre, prospective, placebo-controlled, double-blind, randomized, 3-arm parallel group, interventional study is to assess for the first time the effects of either a combined therapy with the antihyperglycemic drugs semaglutide and empagliflozin or empagliflozin monotherapy compared to placebo as potential treatments for non-alcoholic steatohepatitis (NASH) in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Obesity and type 2 diabetes (T2D) are tightly associated with non-alcoholic fatty liver disease (NAFLD), which in turn predicts the development of T2D and cardiovascular disease.

Up to 80% of NAFLD patients with T2D have NASH and the presence of T2D is an independent risk factor for more-advanced fibrosis, higher rate of fibrosis progression, and increased mortality. Liver-related mortality is increased 10-fold in NASH patients compared with the general population. In addition, people with NASH are at an excessive risk of cardiovascular morbidity and mortality.

Currently, there are no established pharmacotherapies for NASH patients with T2D.

The aim of this trial is to evaluate efficacy of a combined treatment with semaglutide 1 mg/week (GLP1RA) and empagliflozin 10 mg/d (SGLT2I) or ii) empagliflozin 10 mg/d monotherapy by means of histological resolution of NASH in T2D patients without progression of fibrosis after 48 weeks treatment.

To confirm a histological diagnosis of NASH and proof efficacy of treatment, a liver biopsy will be performed prior to screening as well as at the end of treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2D and NASH with fibrosis stage F1-F3
* Age between 25 and 75 years
* HbA1c ≤ 9.5%
* obtained written informed consent

Exclusion Criteria:

* Contraindications on liver biopsy
* Evidence of cirrhosis on liver biopsy
* Liver disease of other etiology including chronic viral hepatitis (B or C), alcohol abuse, hemochromatosis, alpha-1 antitrypsin deficiency, autoimmune hepatitis, Wilson's disease, primary sclerosing cholangitis or primary biliary cirrhosis, or liver cirrhosis of any etiology
* History of ketoacidosis
* Alcohol consumption >30 g/d for males and >20 g/d for females
* Past (≥5 years) or current history of alcohol or drug abuse and/or psychiatric disease including severe depression necessitating pharmacological treatment
* Medications that may induce steatosis:tamoxifen, raloxifene, oral glucocorticoids or chloroquine
* Planned pregnancy, pregnant or lactating women, positive pregnancy test, and woman of childbearing potential not using two adequate methods of contraception, including a barrier method and a highly efficacious non-barrier method

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2021-03-26 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Histological resolution of NASH without worsening of fibrosis | from baseline to 48 weeks
  NAFLD status will be assessed by histologic evaluation of liver biopsy samples based on NAFLD activity score. NASH resolution is defined by disappearance of ballooning (score 0), together with either disappearance of lobular inflammation or the persistence of mild lobular inflammation only (score 0 or 1) and resulting in an overall pathologic diagnosis of either steatosis alone or steatosis with mild inflammation; with no worsening of fibrosis. Worsening of fibrosis is defined by an increase of at least one stage of the Kleiner fibrosis classification.

SECONDARY OUTCOMES:
Overall NAFLD activity score (NAS) | from baseline to 48 weeks
  Sum of a) steatosis (0-3 points), b) lobular inflammation (scored 0-3 points), c) hepatocellular ballooning (scored 0-2 points) assessed by liver histology
Stage of fibrosis according to the Kleiner Fibrosis Classification | from baseline to 48 weeks
  Assessed by liver histology according to the Kleiner Fibrosis Classification (stages 0-4)
Activity component of NASH according to the steatosis-activity-fibrosis (SAF) score | from baseline to 48 weeks
  Sum of lobular inflammation (scored 0-3 points)and hepatocellular ballooning (scored 0-2 points) assessed by liver histology
Hepatic steatosis grade | from baseline to 48 weeks
  steatosis grade (0-3) assessed by liver histology

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Principal Investigator — German Diabetes Center
Locations (25):
- Austria (5):
  - Medizinische Universität Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Wiener Gesundheitsverbund, Klinik Landstraße, Vienna
  - Medizinische Universität Wien, Vienna
  - Wiener Gesundheitsverbund, Klinik Hietzing, Vienna
- Germany (20):
  - German Diabetes Center, Düsseldorf, North Rhine-Westphalia
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Franziskus-Krankenhaus Berlin, Berlin
  - Leber- und Studienzentrum Checkpoint, Berlin
  - University Clinics Berlin Charité, Berlin
  - University Clinics Bochum, Bochum
  - Städtisches Klinikum Brandenburg GmbH, Brandenburg
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - University Clinics Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - University Clinics Essen, Essen
  - University Clinics Frankfurt, Frankfurt
  - University Clinics Freiburg, Freiburg im Breisgau
  - University Clinics Heidelberg, Heidelberg
  - Eugastro GmbH, Leipzig
  - University Clinics Johannes-Gutenberg Mainz, Mainz
  - TUM, München
  - University Clinics Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - University Clinics Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No